CLINICAL TRIAL: NCT03882957
Title: Media Multi-tasking and Cued Overeating: Assessing the Pathway and Piloting an Intervention Using an Attentional Network Framework
Brief Title: Trial on the Effect of Media Multi-tasking on Attention to Food Cues and Cued Overeating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Dartmouth College (Other)
Responsible Party: Principal Investigator, Diane Gilbert-Diamond, Associate Professor of Epidemiology and Community and Family Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: D19065; 1R21HD097475-01 (NIH)
Record Dates: First submitted 2019-03-19; First posted 2019-03-20 (Actual); Results first posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Attention Concentration Difficulty; Obesity, Childhood
Keywords: Attention; Food cues; Media multi-tasking
MeSH Terms: conditions — Pediatric Obesity | interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: This is a within-subject design where each participant is randomly assigned to all three arms.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video (Active Comparator): videos of media tasks being completed
  Interventions: Other: Video
- media multi-task (Experimental): media tasks
  Interventions: Behavioral: media multi-task
- sustained attention task (Experimental): a cognitive task that trains sustained attention
  Interventions: Behavioral: Sustained attention

INTERVENTIONS:
Behavioral: Sustained attention — participants will complete a sustained attention task
  Arms: sustained attention task
Behavioral: media multi-task — participants will complete multiple media tasks at the same time
  Arms: media multi-task
Other: Video — participants will watch a video of media tasks being completed
  Arms: Video

SUMMARY:
Childhood obesity is a critical public health problem in the United States. One factor known to contribute to childhood obesity is excess consumption. Importantly, excess consumption related to weight gain is not necessarily driven by hunger. For example, environmental food cues stimulate brain reward regions and lead to overeating even after a child has eaten to satiety. This type of cued eating is associated with increased attention to food cues; the amount of time a child spends looking at food cues (e.g., food advertisements) is associated with increased caloric intake. However, individual susceptibility to environmental food cues remains unknown. It is proposed that the prevalent practice of media multi-tasking-simultaneously attending to multiple electronic media sources-increases attention to peripheral food cues in the environment and thereby plays an important role in the development of obesity. It is hypothesized that multi-tasking teaches children to engage in constant task switching that makes them more responsive to peripheral cues, many of which are potentially harmful (such as those that promote overeating). The overarching hypothesis is that media multi-tasking alters the attentional networks of the brain that control attention to environmental cues. High media multi-tasking children are therefore particularly susceptible to food cues, thereby leading to increased cued eating. It is also predicted that attention modification training can provide a protective effect against detrimental attentional processing caused multi-tasking, by increasing the proficiency of the attention networks. These hypotheses will be tested by assessing the pathway between media-multitasking, attention to food cues, and cued eating. It will also be examined whether it is possible to intervene on this pathway by piloting an at-home attention modification training intervention designed to reduce attention to food cues. It is our belief that this research will lead to the development of low-cost, scalable tools that can train attention networks so that children are less influenced by peripheral food cues, a known cause of overeating. For example, having children practice attention modification intervention tasks regularly (which could be accomplished through user-friendly computer games or cell phone/tablet apps) might offset the negative attentional effects of media multi-tasking.

DETAILED DESCRIPTION:
[3/14/2020]: Study recruitment temporarily halted due to the COVID-19 pandemic

ELIGIBILITY:
Inclusion Criteria:

* N/A.

Exclusion Criteria:

* Inadequate English proficiency, a vision disorder that is not corrected with corrective lenses, and relevant food allergies.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Gilbert-Diamond, ScD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth-Hithchock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rapuano KM, Zieselman AL, Kelley WM, Sargent JD, Heatherton TF, Gilbert-Diamond D. Genetic risk for obesity predicts nucleus accumbens size and responsivity to real-world food cues. Proc Natl Acad Sci U S A. 2017 Jan 3;114(1):160-165. doi: 10.1073/pnas.1605548113. Epub 2016 Dec 19. PMID 27994159
- [Background] Folkvord F, Anschutz DJ, Wiers RW, Buijzen M. The role of attentional bias in the effect of food advertising on actual food intake among children. Appetite. 2015 Jan;84:251-8. doi: 10.1016/j.appet.2014.10.016. Epub 2014 Oct 22. PMID 25451582
- [Background] Corbetta M, Patel G, Shulman GL. The reorienting system of the human brain: from environment to theory of mind. Neuron. 2008 May 8;58(3):306-24. doi: 10.1016/j.neuron.2008.04.017. PMID 18466742
- [Background] Corbetta M, Shulman GL. Control of goal-directed and stimulus-driven attention in the brain. Nat Rev Neurosci. 2002 Mar;3(3):201-15. doi: 10.1038/nrn755. PMID 11994752
- [Background] Hou Y, Liu T. Neural correlates of object-based attentional selection in human cortex. Neuropsychologia. 2012 Oct;50(12):2916-2925. doi: 10.1016/j.neuropsychologia.2012.08.022. Epub 2012 Sep 4. PMID 22963835
- [Background] Moisala M, Salmela V, Hietajarvi L, Salo E, Carlson S, Salonen O, Lonka K, Hakkarainen K, Salmela-Aro K, Alho K. Media multitasking is associated with distractibility and increased prefrontal activity in adolescents and young adults. Neuroimage. 2016 Jul 1;134:113-121. doi: 10.1016/j.neuroimage.2016.04.011. Epub 2016 Apr 8. PMID 27063068
- [Background] Yap JY, Lim SWH. Media multitasking predicts unitary versus splitting visual focal attention. Journal of Cognitive Psychology. Routledge; 2013 Nov;25(7):889-902.
- [Background] Ophir E, Nass C, Wagner AD. Cognitive control in media multitaskers. Proc Natl Acad Sci U S A. 2009 Sep 15;106(37):15583-7. doi: 10.1073/pnas.0903620106. Epub 2009 Aug 24. PMID 19706386
- [Background] Boutelle KN, Kuckertz JM, Carlson J, Amir N. A pilot study evaluating a one-session attention modification training to decrease overeating in obese children. Appetite. 2014 May;76:180-5. doi: 10.1016/j.appet.2014.01.075. Epub 2014 Feb 8. PMID 24512975
- [Background] Posner MI, Petersen SE. The attention system of the human brain. Annu Rev Neurosci. 1990;13:25-42. doi: 10.1146/annurev.ne.13.030190.000325. No abstract available. PMID 2183676
- [Background] Pozuelos JP, Paz-Alonso PM, Castillo A, Fuentes LJ, Rueda MR. Development of attention networks and their interactions in childhood. Dev Psychol. 2014 Oct;50(10):2405-15. doi: 10.1037/a0037469. Epub 2014 Jul 28. PMID 25069052
- [Background] Hill LJ, Coats RO, Mushtaq F, Williams JH, Aucott LS, Mon-Williams M. Moving to Capture Children's Attention: Developing a Methodology for Measuring Visuomotor Attention. PLoS One. 2016 Jul 19;11(7):e0159543. doi: 10.1371/journal.pone.0159543. eCollection 2016. PMID 27434198
- [Background] Birch LL, Fisher JO. Development of eating behaviors among children and adolescents. Pediatrics. 1998 Mar;101(3 Pt 2):539-49. PMID 12224660
- [Background] Rideout VJ, Foehr UG, Roberts DF. Generation M2: Media in the lives of 8- to 10-year olds. 2010 Jan.
- [Background] Rideout VJ. Zero to eight: Children's media use in America 2013. New York, New York: Common Sense Media.
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Han JC, Lawlor DA, Kimm SY. Childhood obesity. Lancet. 2010 May 15;375(9727):1737-48. doi: 10.1016/S0140-6736(10)60171-7. Epub 2010 May 5. PMID 20451244
- [Background] Daniels SR, Arnett DK, Eckel RH, Gidding SS, Hayman LL, Kumanyika S, Robinson TN, Scott BJ, St Jeor S, Williams CL. Overweight in children and adolescents: pathophysiology, consequences, prevention, and treatment. Circulation. 2005 Apr 19;111(15):1999-2012. doi: 10.1161/01.CIR.0000161369.71722.10. PMID 15837955
- [Background] Biro FM, Wien M. Childhood obesity and adult morbidities. Am J Clin Nutr. 2010 May;91(5):1499S-1505S. doi: 10.3945/ajcn.2010.28701B. Epub 2010 Mar 24. PMID 20335542
- [Background] Whitaker RC, Wright JA, Pepe MS, Seidel KD, Dietz WH. Predicting obesity in young adulthood from childhood and parental obesity. N Engl J Med. 1997 Sep 25;337(13):869-73. doi: 10.1056/NEJM199709253371301. PMID 9302300
- [Background] Serdula MK, Ivery D, Coates RJ, Freedman DS, Williamson DF, Byers T. Do obese children become obese adults? A review of the literature. Prev Med. 1993 Mar;22(2):167-77. doi: 10.1006/pmed.1993.1014. PMID 8483856
- [Background] Guyenet SJ, Schwartz MW. Clinical review: Regulation of food intake, energy balance, and body fat mass: implications for the pathogenesis and treatment of obesity. J Clin Endocrinol Metab. 2012 Mar;97(3):745-55. doi: 10.1210/jc.2011-2525. Epub 2012 Jan 11. PMID 22238401
- [Background] Lutter M, Nestler EJ. Homeostatic and hedonic signals interact in the regulation of food intake. J Nutr. 2009 Mar;139(3):629-32. doi: 10.3945/jn.108.097618. Epub 2009 Jan 28. PMID 19176746
- [Background] Boswell RG, Kober H. Food cue reactivity and craving predict eating and weight gain: a meta-analytic review. Obes Rev. 2016 Feb;17(2):159-77. doi: 10.1111/obr.12354. Epub 2015 Dec 8. PMID 26644270
- [Background] Demos KE, Heatherton TF, Kelley WM. Individual differences in nucleus accumbens activity to food and sexual images predict weight gain and sexual behavior. J Neurosci. 2012 Apr 18;32(16):5549-52. doi: 10.1523/JNEUROSCI.5958-11.2012. PMID 22514316
- [Background] Davids S, Lauffer H, Thoms K, Jagdhuhn M, Hirschfeld H, Domin M, Hamm A, Lotze M. Increased dorsolateral prefrontal cortex activation in obese children during observation of food stimuli. Int J Obes (Lond). 2010 Jan;34(1):94-104. doi: 10.1038/ijo.2009.193. Epub 2009 Oct 6. PMID 19806158
- [Background] Bruce AS, Holsen LM, Chambers RJ, Martin LE, Brooks WM, Zarcone JR, Butler MG, Savage CR. Obese children show hyperactivation to food pictures in brain networks linked to motivation, reward and cognitive control. Int J Obes (Lond). 2010 Oct;34(10):1494-500. doi: 10.1038/ijo.2010.84. Epub 2010 May 4. PMID 20440296
- [Background] Lawrence NS, Hinton EC, Parkinson JA, Lawrence AD. Nucleus accumbens response to food cues predicts subsequent snack consumption in women and increased body mass index in those with reduced self-control. Neuroimage. 2012 Oct 15;63(1):415-22. doi: 10.1016/j.neuroimage.2012.06.070. Epub 2012 Jul 6. PMID 22776461
- [Background] Hill JO, Peters JC. Environmental contributions to the obesity epidemic. Science. 1998 May 29;280(5368):1371-4. doi: 10.1126/science.280.5368.1371. PMID 9603719
- [Background] Rodearmel SJ, Wyatt HR, Stroebele N, Smith SM, Ogden LG, Hill JO. Small changes in dietary sugar and physical activity as an approach to preventing excessive weight gain: the America on the Move family study. Pediatrics. 2007 Oct;120(4):e869-79. doi: 10.1542/peds.2006-2927. PMID 17908743
- [Background] Castellanos EH, Charboneau E, Dietrich MS, Park S, Bradley BP, Mogg K, Cowan RL. Obese adults have visual attention bias for food cue images: evidence for altered reward system function. Int J Obes (Lond). 2009 Sep;33(9):1063-73. doi: 10.1038/ijo.2009.138. Epub 2009 Jul 21. PMID 19621020
- [Background] Yager LM, Robinson TE. Cue-induced reinstatement of food seeking in rats that differ in their propensity to attribute incentive salience to food cues. Behav Brain Res. 2010 Dec 6;214(1):30-4. doi: 10.1016/j.bbr.2010.04.021. Epub 2010 Apr 21. PMID 20416342
- [Background] Hickey C, Peelen MV. Neural mechanisms of incentive salience in naturalistic human vision. Neuron. 2015 Feb 4;85(3):512-8. doi: 10.1016/j.neuron.2014.12.049. PMID 25654257
- [Background] Brockmeyer T, Hahn C, Reetz C, Schmidt U, Friederich HC. Approach bias and cue reactivity towards food in people with high versus low levels of food craving. Appetite. 2015 Dec;95:197-202. doi: 10.1016/j.appet.2015.07.013. Epub 2015 Jul 13. PMID 26184338
- [Background] Hendrikse JJ, Cachia RL, Kothe EJ, McPhie S, Skouteris H, Hayden MJ. Attentional biases for food cues in overweight and individuals with obesity: a systematic review of the literature. Obes Rev. 2015 May;16(5):424-32. doi: 10.1111/obr.12265. Epub 2015 Mar 5. PMID 25752592
- [Background] Kemps E, Tiggemann M, Orr J, Grear J. Attentional retraining can reduce chocolate consumption. J Exp Psychol Appl. 2014 Mar;20(1):94-102. doi: 10.1037/xap0000005. Epub 2013 Sep 30. PMID 24079387
- [Background] Jha AP, Krompinger J, Baime MJ. Mindfulness training modifies subsystems of attention. Cogn Affect Behav Neurosci. 2007 Jun;7(2):109-19. doi: 10.3758/cabn.7.2.109. PMID 17672382
- [Background] Hardman CA, Rogers PJ, Etchells KA, Houstoun KV, Munafo MR. The effects of food-related attentional bias training on appetite and food intake. Appetite. 2013 Dec;71:295-300. doi: 10.1016/j.appet.2013.08.021. Epub 2013 Sep 8. PMID 24025548
- [Background] Kleiman T, Trope Y, Amodio DM. Cognitive control modulates attention to food cues: Support for the control readiness model of self-control. Brain Cogn. 2016 Dec;110:94-101. doi: 10.1016/j.bandc.2016.04.006. Epub 2016 May 3. PMID 27157690
- [Background] Amir N, Weber G, Beard C, Bomyea J, Taylor CT. The effect of a single-session attention modification program on response to a public-speaking challenge in socially anxious individuals. J Abnorm Psychol. 2008 Nov;117(4):860-868. doi: 10.1037/a0013445. PMID 19025232
- [Background] Sturm W, Thimm M, Kust J, Karbe H, Fink GR. Alertness-training in neglect: behavioral and imaging results. Restor Neurol Neurosci. 2006;24(4-6):371-84. PMID 17119311
- [Background] Thimm M, Fink GR, Kust J, Karbe H, Sturm W. Impact of alertness training on spatial neglect: a behavioural and fMRI study. Neuropsychologia. 2006;44(7):1230-46. doi: 10.1016/j.neuropsychologia.2005.09.008. Epub 2005 Nov 8. PMID 16280140
- [Background] Gorman TE, Green CS. Short-term mindfulness intervention reduces the negative attentional effects associated with heavy media multitasking. Sci Rep. 2016 Apr 18;6:24542. doi: 10.1038/srep24542. PMID 27086504
- [Background] Robertson IH, Manly T, Andrade J, Baddeley BT, Yiend J. 'Oops!': performance correlates of everyday attentional failures in traumatic brain injured and normal subjects. Neuropsychologia. 1997 Jun;35(6):747-58. doi: 10.1016/s0028-3932(97)00015-8. PMID 9204482
- [Background] Mrazek MD, Smallwood J, Schooler JW. Mindfulness and mind-wandering: finding convergence through opposing constructs. Emotion. 2012 Jun;12(3):442-448. doi: 10.1037/a0026678. Epub 2012 Feb 6. PMID 22309719
- [Background] Rueda MR, Fan J, McCandliss BD, Halparin JD, Gruber DB, Lercari LP, Posner MI. Development of attentional networks in childhood. Neuropsychologia. 2004;42(8):1029-40. doi: 10.1016/j.neuropsychologia.2003.12.012. PMID 15093142
- [Background] Federico F, Marotta A, Martella D, Casagrande M. Development in attention functions and social processing: Evidence from the Attention Network Test. Br J Dev Psychol. 2017 Jun;35(2):169-185. doi: 10.1111/bjdp.12154. Epub 2016 Aug 4. PMID 27491798
- [Background] Gilbert-Diamond D, Emond JA, Lansigan RK, Rapuano KM, Kelley WM, Heatherton TF, Sargent JD. Television food advertisement exposure and FTO rs9939609 genotype in relation to excess consumption in children. Int J Obes (Lond). 2017 Jan;41(1):23-29. doi: 10.1038/ijo.2016.163. Epub 2016 Sep 22. PMID 27654143
- [Background] Emond JA, Lansigan RK, Ramanujam A, Gilbert-Diamond D. Randomized Exposure to Food Advertisements and Eating in the Absence of Hunger Among Preschoolers. Pediatrics. 2016 Dec;138(6):e20162361. doi: 10.1542/peds.2016-2361. PMID 27940713
- [Background] Hill C, Llewellyn CH, Saxton J, Webber L, Semmler C, Carnell S, van Jaarsveld CH, Boniface D, Wardle J. Adiposity and 'eating in the absence of hunger' in children. Int J Obes (Lond). 2008 Oct;32(10):1499-505. doi: 10.1038/ijo.2008.113. Epub 2008 Jul 22. PMID 18645573
- [Background] Heatherton TF, Wagner DD. Cognitive neuroscience of self-regulation failure. Trends Cogn Sci. 2011 Mar;15(3):132-9. doi: 10.1016/j.tics.2010.12.005. Epub 2011 Jan 26. PMID 21273114
- [Background] Wagner DD, Altman M, Boswell RG, Kelley WM, Heatherton TF. Self-regulatory depletion enhances neural responses to rewards and impairs top-down control. Psychol Sci. 2013 Nov 1;24(11):2262-71. doi: 10.1177/0956797613492985. Epub 2013 Sep 11. PMID 24026225
- [Background] Wagner DD, Boswell RG, Kelley WM, Heatherton TF. Inducing negative affect increases the reward value of appetizing foods in dieters. J Cogn Neurosci. 2012 Jul;24(7):1625-33. doi: 10.1162/jocn_a_00238. Epub 2012 Apr 23. PMID 22524295
- [Background] Petersen SE, Posner MI. The attention system of the human brain: 20 years after. Annu Rev Neurosci. 2012;35:73-89. doi: 10.1146/annurev-neuro-062111-150525. Epub 2012 Apr 12. PMID 22524787
- [Background] Duc AH, Bays P, Husain M. Eye movements as a probe of attention. Prog Brain Res. 2008;171:403-11. doi: 10.1016/S0079-6123(08)00659-6. PMID 18718333
- [Background] Armstrong T, Olatunji BO. Eye tracking of attention in the affective disorders: a meta-analytic review and synthesis. Clin Psychol Rev. 2012 Dec;32(8):704-23. doi: 10.1016/j.cpr.2012.09.004. Epub 2012 Sep 20. PMID 23059623
- [Background] Adler SA, Gallego P. Search asymmetry and eye movements in infants and adults. Atten Percept Psychophys. 2014 Aug;76(6):1590-608. doi: 10.3758/s13414-014-0667-6. PMID 24858309
- [Background] Fisher JO, Birch LL. Eating in the absence of hunger and overweight in girls from 5 to 7 y of age. Am J Clin Nutr. 2002 Jul;76(1):226-31. doi: 10.1093/ajcn/76.1.226. PMID 12081839
- [Background] Alzahabi R, Becker MW. The association between media multitasking, task-switching, and dual-task performance. J Exp Psychol Hum Percept Perform. 2013 Oct;39(5):1485-1495. doi: 10.1037/a0031208. Epub 2013 Feb 11. PMID 23398256
- [Background] Ralph BC, Thomson DR, Seli P, Carriere JS, Smilek D. Media multitasking and behavioral measures of sustained attention. Atten Percept Psychophys. 2015 Feb;77(2):390-401. doi: 10.3758/s13414-014-0771-7. PMID 25280520
- [Background] Hillman CH, Pontifex MB, Raine LB, Castelli DM, Hall EE, Kramer AF. The effect of acute treadmill walking on cognitive control and academic achievement in preadolescent children. Neuroscience. 2009 Mar 31;159(3):1044-54. doi: 10.1016/j.neuroscience.2009.01.057. Epub 2009 Feb 3. PMID 19356688
- [Background] LeBlanc AG, Katzmarzyk PT, Barreira TV, Broyles ST, Chaput JP, Church TS, Fogelholm M, Harrington DM, Hu G, Kuriyan R, Kurpad A, Lambert EV, Maher C, Maia J, Matsudo V, Olds T, Onywera V, Sarmiento OL, Standage M, Tudor-Locke C, Zhao P, Tremblay MS; ISCOLE Research Group. Correlates of Total Sedentary Time and Screen Time in 9-11 Year-Old Children around the World: The International Study of Childhood Obesity, Lifestyle and the Environment. PLoS One. 2015 Jun 11;10(6):e0129622. doi: 10.1371/journal.pone.0129622. eCollection 2015. PMID 26068231
- [Background] Katzmarzyk PT, Barreira TV, Broyles ST, Champagne CM, Chaput JP, Fogelholm M, Hu G, Johnson WD, Kuriyan R, Kurpad A, Lambert EV, Maher C, Maia J, Matsudo V, Olds T, Onywera V, Sarmiento OL, Standage M, Tremblay MS, Tudor-Locke C, Zhao P, Church TS. The International Study of Childhood Obesity, Lifestyle and the Environment (ISCOLE): design and methods. BMC Public Health. 2013 Sep 30;13:900. doi: 10.1186/1471-2458-13-900. PMID 24079373
- [Background] Mitchell JA, Pate RR, Beets MW, Nader PR. Time spent in sedentary behavior and changes in childhood BMI: a longitudinal study from ages 9 to 15 years. Int J Obes (Lond). 2013 Jan;37(1):54-60. doi: 10.1038/ijo.2012.41. Epub 2012 Mar 20. PMID 22430304
- [Background] Petersen AC, Crockett L, Richards M, Boxer A. A self-report measure of pubertal status: Reliability, validity, and initial norms. J Youth Adolesc. 1988 Apr;17(2):117-33. doi: 10.1007/BF01537962. PMID 24277579
- [Background] Carskadon MA, Acebo C. A self-administered rating scale for pubertal development. J Adolesc Health. 1993 May;14(3):190-5. doi: 10.1016/1054-139x(93)90004-9. PMID 8323929
- [Background] Brooks-Gunn J, Warren MP, Rosso J, Gargiulo J. Validity of self-report measures of girls' pubertal status. Child Dev. 1987 Jun;58(3):829-41. PMID 3608653
- [Background] Dixon HG, Scully ML, Wakefield MA, White VM, Crawford DA. The effects of television advertisements for junk food versus nutritious food on children's food attitudes and preferences. Soc Sci Med. 2007 Oct;65(7):1311-23. doi: 10.1016/j.socscimed.2007.05.011. Epub 2007 Jun 22. PMID 17587474
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319
- [Background] Marshall TA, Eichenberger Gilmore JM, Broffitt B, Stumbo PJ, Levy SM. Relative validity of the Iowa Fluoride Study targeted nutrient semi-quantitative questionnaire and the block kids' food questionnaire for estimating beverage, calcium, and vitamin D intakes by children. J Am Diet Assoc. 2008 Mar;108(3):465-72. doi: 10.1016/j.jada.2007.12.002. PMID 18313429
- [Background] Wardle J, Guthrie CA, Sanderson S, Rapoport L. Development of the Children's Eating Behaviour Questionnaire. J Child Psychol Psychiatry. 2001 Oct;42(7):963-70. doi: 10.1111/1469-7610.00792. PMID 11693591
- [Background] Lohman TG, Roche AF, Martorell R. Anthropometric standardization reference manual. Champaign Ill: Human Kinetics Books; 1991.
- [Background] CDC growth charts: United States [Internet]. Washington, DC. Available from: http://www.cdc.gov.growthcharts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 92 Adolescents were enrolled in this study.
Groups:
- All Study Participants: This study has a within-subject design where each participant is assigned to all three arms in a randomized manner. The various sequences were:
  video --> media multitask --> sustained attention video --> sustained attention --> media multitask media multitask --> video --> sustained attention sustained attention --> video --> media multitask sustained attention --> media multitask --> video media multitask --> sustained attention --> video
Period: Overall Study
Arm/Group | All Study Participants
Started | 92
Participant Flow 1 | 17 (participant flow sequence: video --> media multitask --> sustained attention)
Participant Flow 2 | 16 (participant flow sequence: video --> sustained attention -- media multitask)
Participant Flow 3 | 13 (participant flow sequence: media multitask --> video --> sustained attention)
Participant Flow 4 | 15 (participant flow sequence: sustained attention --> video -- media multitask)
Participant Flow 5 | 16 (participant flow sequence: sustained attention --> media multitask --> video)
Participant Flow 6 | 14 (participant flow 6: media multitask --> sustained attention --> video)
Completed | 91
Not Completed | 1
Not completed — Did not complete all three arms | 1

BASELINE CHARACTERISTICS:
Groups:
- Individual Participant Data.: This study has a within-subject design where each participant is assigned to all three arms in a randomized fashion. Baseline population data was only collected for adolescents.
Arm/Group | Individual Participant Data.
Number analyzed (Participants) | 92
Age, Customized [Count of Participants; unit: Participants]
  Age 13 | 24
  Age 14 | 23
  Age 15 | 26
  Age 16 | 15
  Age 17 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 87
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 80
  More than one race | 5
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 92

OUTCOME MEASURES:

1. Primary Outcome: Amount of Time Spent Looking at Food Cues While Playing a Media Game
Description: Eye-tracking will be used to measure the amount of time spent looking at static food cues while participants play a media game on the computer. The amount time spent looking at a food cue is a measure how much attention was given to the food cue. The longer the looking time, the greater amount of attention.
Time Frame: approximately 15 minutes post-intervention
Population: Cumulative fixation duration. Five children were excluded from the computation of these eye tracking metric because of unsuccessful eye tracking calibration.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Video (Control): videos of media tasks being completed
  Video: participants will watch a video of media tasks being completed
Arm/Group | Video (Control) | Media Multi-task | Sustained Attention Task
Number analyzed (Participants) | 86 | 86 | 86
milliseconds
  Animals (control) | 9304.26 (15332.66) | 10196.45 (12806.60) | 8654.48 (14717.66)
  Food | 8486.79 (13977.62) | 11367.48 (13858.05) | 8802.22 (13605.90)
  Total | 17791.05 (23852.25) | 21563.93 (21466.33) | 17662.07 (22825.76)

2. Primary Outcome: Amount of Snack Foods Consumed Post-intervention
Description: The amount of kcals consumed of snack foods after participants have completed the intervention.
Time Frame: approximately 30 minutes post-intervention
Population: A single participant dropped out after completing 2 visits, failing to complete their control condition visit.
Measure: Mean (Standard Deviation); unit: kcals
Arm/Group | Video (Control) | Media Multi-task | Sustained Attention Task
Number analyzed (Participants) | 91 | 92 | 92
kcals | 435.18 (208.76) | 423.99 (183.32) | 433.54 (185.22)

3. Primary Outcome: Daily Usual Media Multi-tasking
Description: Participants reported on their usual media multitasking using the short form media multitasking index. This index asks about media multitasking with other print and digital media during four primary activities: 1) watching television or movies, 2) playing video games, 3) reading books or magazines (not assigned for school), and 4) doing homework. For each activity, participants reported the frequency with which they multitasked by engaging in the other activities by using a 5-point likert scale (i.e., 0=Never, 1=Rarely, 2=Sometimes, 3=Often, 4=Always). A usual media multitasking score was computed by taking the average of the Likert response. The score ranges from 0 to 4 with a higher score indicative of higher self-reported usual media multitasking.
Time Frame: approximately 10 minutes prior to the intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Media Multitasking Scores
Number analyzed (Participants) | 91
units on a scale | 2.35 (0.87)

ADVERSE EVENTS:
Time Frame: This study did not track adverse events.
Description: This study did not track adverse events.
Arm/Group | Video | Media Multi-task | Sustained Attention Task
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT03882957/Prot_SAP_002.pdf
  • Informed Consent Form: Informed Consent Form: Adult (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT03882957/ICF_000.pdf
  • Informed Consent Form: Informed Assent Form: Child (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT03882957/ICF_001.pdf